CLINICAL TRIAL: NCT06942182
Title: Double Blind Placebo-Controlled Parallel Group Study Of Safety And Efficacy Of Isomyosamine In Treating Sarcopenia After Hip Or Femoral Fracture In Gerontological Population
Brief Title: Safety and Efficacy of Isomyosamine in Reducing Inflammation and Treating Muscle Loss in Older Adults After Hip or Thigh Bone Fractures
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TNF Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNF001
Record Dates: First submitted 2025-04-09; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Sarcopenia in Elderly; Frailty; Frailty/Sarcopenia; Frailty in Older Adults
Keywords: sarcopenia; Frailty; Hip Fracture; Older population; Gerontological; Femur fracture; Sarcopenia and Frailty
MeSH Terms: conditions — Frailty; Sarcopenia; Hip Fractures; Femoral Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Drug: 1000 mg Isomyosamine (Experimental): Subjects randomly assigned to receive 1000 mg Isomyosamine daily via four 250 mg capsules
  Interventions: Drug: Isomyosamine 250mg
- Placebo 1000 mg (Placebo Comparator): Subjects randomly assigned to receive 1000 mg placebo daily via four 250 mg capsules
  Interventions: Drug: Placebo 250 mg

INTERVENTIONS:
Drug: Isomyosamine 250mg — Isomyosamine 250 mg capsules dosed 4 times daily
  Arms: Study Drug: 1000 mg Isomyosamine
Drug: Placebo 250 mg — Placebo 250 mg capsule 4 times daily
  Arms: Placebo 1000 mg

SUMMARY:
This Phase II clinical study investigates the safety and effectiveness of a new drug, Isomyosamine, in patients with sarcopenia or frailty, conditions associated with aging and muscle weakness. Isomyosamine is a promising oral medication that reduces inflammation by targeting cytokines like TNF-α and IL-6, which are linked to these conditions. Previous studies have shown it is well-tolerated and may help improve muscle strength, mobility, and healing after hip fractures. This trial aims to determine its potential benefits in reducing inflammation and improving recovery in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 to 85 years of age
2. Non-complex, non-comminuted fracture of the femoral head, femoral neck, or acetabulum due to an accidental (non-neurologic or cardiovascular) fall
3. Concomitant medication limited to treatment for chronic conditions
4. The ability to give informed consent and comply with study procedures
5. Body weight ≥35 kg
6. Adequate dietary intake
7. Potential subjects' intention to avoid reproductive activity will be confirmed

   And one or more of the following criteria:
8. Previous history frailty or sarcopenia diagnosis using standardized tests;
9. Positive assessment for frailty or sarcopenia using standardized tests or as per clinician's judgement;
10. Previous positive assessment for elevated biomarkers of inflammation (serum IL-6 level> LOQ, TNFR1 level > LOQ, and/or TNF-alpha level > LOQ)

Exclusion Criteria:

1. Receiving immunotherapy for cancer or solid organ transplantation
2. Complex or comminuted fracture or fracture of multiple long bones
3. Regular treatment for chronic disease including chronic renal failure, chronic heart failure (CHF) cerebrovascular disease including stroke, rheumatoid arthritis, or polymyalgia rheumatica
4. Chronic kidney disease (estimated glomerular filtration rate [eGFR] <60 mL/min)
5. Newly (< 2 weeks) diagnosed COVID-19
6. Inability or unwillingness to give written informed consent
7. History of upper/lower respiratory tract infection, requiring systemic steroids, antibiotics, and or emergency room (ER) visit or urgent care within 6 weeks of screening visit
8. History of adverse reaction or allergy to TNF inhibitor
9. History of neurological, hepatic, renal, diabetic mellitus, thyroid disorder, psychiatric, addiction or other medical conditions that may interfere with the interpretation of data or the patient's participation in the study or may increase safety concerns per investigator discretion
10. Currently under treatment by an anti-TNFα drug, such as adalimumab, etanercept, infliximab, certolizumab pegol, golimumab, and biosimilars
11. Currently under treatment by an anti-diabetic medication, including glucagon-like peptide-1 (GLP-1) drugs such as semaglutide, or any of metformin, jenuvia, or insulin
12. Unwillingness or inability to comply with study procedures, including smoking cessation
13. History of epilepsy or seizure propensity, ataxia, abnormal EEG findings, abnormal brain magnetic resonance image, or other co-morbid neurological conditions
14. Positive TB test
15. Patients who are pregnant or breastfeeding

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) Test in subjects treated with Isomyosamine or placebo | From enrollment to the end of treatment at 90 days

SECONDARY OUTCOMES:
4-meter walk test | From enrollment to the end of treatment at 90 days
  Change in the time taken to walk 4 meters through 90 days dosing.
6-minute walk test | From enrollment to the end of treatment at 90 days
  Change in the distance walked in the 6-minute walk test (m) through 90 days dosing.
Grip strength | From enrollment to the end of treatment at 90 days
  Change in grip strength score over 90 day dosing.
Effect on serum levels of biochemical markers of TNF activation | From enrollment to the end of treatment at 90 days
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 in the Isomyosamine vs Placebo groups | From enrollment to the end of treatment at 90 days

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://tnfpharma.com/